CLINICAL TRIAL: NCT05868356
Title: A Phase 1, Open-label, Multiple-dose, One-sequence Crossover Study to Investigate the Effect of Repeated Oral Doses of a Strong CYP2C8 Inhibitor on the Steady-state Pharmacokinetics of Adagrasib in Healthy Adult Subjects
Brief Title: A PK Study to Assess the Drug-drug Interaction of a Strong CYP2C8 Inhibitor on Adagrasib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 849-024
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: A Phase 1, Open-label, Multiple-dose, One-sequence Crossover Study to Investigate the Effect of Repeated Oral Doses of a Strong CYP2C8 Inhibitor on the Steady-state Pharmacokinetics of Adagrasib in Healthy Adult Subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Treatment A — Oral adagrasib 200 mg twice daily (BID) for 8 days (Days 1 to 8). Predose PK blood samples for the measurement of adagrasib concentration will be collected on Days 2 to 7. Serial PK blood samples for adagrasib will be collected up to 12 hours postdose on Days 1 and 8.
Drug: Treatment B — Oral adagrasib 200 mg BID and gemfibrozil 600 mg BID for 10 days (Days 9 to 18), with no evening dose of adagrasib or gemfibrozil on Day 18. Predose PK blood samples for the measurement of adagrasib concentration will be collected on Days 9 to 17 before the morning dose of adagrasib. Predose PK blood samples for the measurement of gemfibrozil trough concentration will be collected on Days 15 to 18 before the morning dose of gemfibrozil. Serial PK blood samples for adagrasib will be collected up to 12 hours postdose on Day 18.

SUMMARY:
A Phase 1, Open-label, Multiple-dose, One-sequence Crossover Study to Investigate the Effect of Repeated Oral Doses of a Strong CYP2C8 Inhibitor on the Steady-state Pharmacokinetics of Adagrasib in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 60 years of age, inclusive, at Screening.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive, at Screening.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, or clinical laboratory evaluations at Screening and Check-in as assessed by the Investigator.
4. Females of childbearing potential will not be pregnant or lactating and must have a negative result on an approved pregnancy test at Screening and Check-in. Females of childbearing potential must agree to use contraception.
5. Male subjects must agree to use contraception.
6. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator.
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, any components of the investigational product (IP), or other substance (not including seasonal allergies).
3. History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions (eg, uncontrolled nausea, vomiting, malabsorption syndrome) likely to alter absorption of study treatment or result in inability to swallow oral medications.
4. Significant history or clinical manifestation of any hepatic disease.
5. History or current diagnosis of uncontrolled or significant cardiac disease.
6. Ventricular dysfunction or history of risk factors for Torsades de Pointes.
7. History of allergic reaction to fibric acid derivatives.
8. History of drug abuse within 2 years prior to Screening.
9. History of alcohol abuse within 12 months prior to Screening.
10. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in.
11. Use of any drugs or substances known or suspected to alter drug absorption, distribution, metabolism, or elimination.
12. Use or intend to use any prescription medications/products within 14 days prior to Check-in.
13. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations.
14. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to Check-in.
15. Participation in a clinical study involving administration of an investigational drug in the past 30 days or 5 half-lives prior to dosing, whichever is longer.
16. Have previously completed or withdrawn from this study or any other study investigating adagrasib, and have previously received the IP.
17. Receipt of blood products within 3 months prior to Check-in.
18. Donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
19. Subjects who, in the opinion of the Investigator, should not participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - AUC (adagrasib) | Days 1, 8, and 18
  Area under the plasma concentration time curve (AUC) during a dosage interval (AUCtau)
Pharmacokinetics - Cmax (adagrasib) | Days 1, 8, and 18
  Maximum observed plasma concentration
Pharmacokinetics - Tmax (adagrasib) | Days 1, 8, and 18
  Time to reach Cmax (tmax)

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to 9 weeks from screening
  Incidence and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Clinical Research Unit Inc, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No